CLINICAL TRIAL: NCT06831630
Title: Comparing the Effects of Holmich Protocol Exercise Therapy and Joint Mobilization Training on Pain, Balance, Function of the Lower Limb, and Muscle Activity in Soccer Players with Athletic Groin Pain.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yeditepe University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Farzadyeditepe
Record Dates: First submitted 2025-02-12; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-01

CONDITIONS: Groin Pain
Keywords: Holmich protocol; Groin Pain; joint mobilization training; Electromyography; pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Holmich protocol exercise (Experimental)
  Interventions: Other: Holmich protocol exercise
- Joint Mobilization (Experimental)
  Interventions: Other: Joint Mobilization
- control (No Intervention)

INTERVENTIONS:
Other: Holmich protocol exercise — The treatment consisted of exercise therapy (ET) protocol suggested by Holmich et al and was started under the supervision of a trained sport physiotherapist who ensured that the exercise was carried out correctly and adhered to the original protocol. No treatment other than ET was applied. Although the ET protocol exactly mirrored the randomised clinical trial of Holmich et al, details such as the perceived resistance or weights (in exercise 3 in module 2) and the rest period between the exercise sets and repetitions, which were not defined in the Holmich study, were explained here for the athletes' benefit (tables 1 and 2). Treatment was administered three times a week (on even or odd days). The duration of each session was about 90 min for module 1 (first two weeks) and 120 min for module 2 (from the third week). From the third week, the athletes were asked to perform exercises from module 1 every other day, between the treatment sessions. Although adductor muscle stretching was for
  Arms: Holmich protocol exercise
Other: Joint Mobilization — Focus of treatment was on reducing hip joint pain using joint mobilization techniques provided by the physical therapist and exercises performed in the HEP. Based on published literature, we developed a standard set of mobilizations to target hip joint motion limitations, defined as stiffness or pain that limited joint range of motion. Joint mobilization techniques were prioritized based on patient-specific tasks and the motion used during those tasks, followed by the hip motion limitations. The choice of joint mobilization techniques and grade used was based on direction of hip motion limitation and the relationship of pain and stiffness during hip motion assessment. The HEP included commonly used joint motion and stretching exercises to complement techniques performed during supervised sessions.
  The exercises will be conducted over a period of 12 weeks, which is explained below Techniques will be prioritized based on restrictions noted on baseline examination.
  1. Caudal glide
  2. Lat
  Arms: Joint Mobilization

SUMMARY:
The goal of this clinical trial is comparison the Holmich protocol exercise therapy and joint mobilization training, investigating their respective effects on muscle activity in soccer players with athletic groin pain.

The main questions it aims to answer are:

Is there a difference between Holmich protocol exercise therapy and joint mobilization training on pain, balance, function of the lower limb, and Muscle activity in Soccer Players with athletic Groin Pain ?

Researchers will compare Holmich protocol exercise therapy (HT)with joint mobilization training (JMT) to see if the exercises are effective on pain, balance, lower limb function, and muscle activity.

Participants will:

Practice Holmich protocol exercise therapy (HT) three times a week, 90 minutes per session, for 12 weeks.

Practice joint mobilization training (JMT) for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male
2. between 18-35 years old
3. Have a normal body mass index (BMI)
4. Desire to return to the former level of sports activity
5. groin pain for at least 2 months
6. Pain at palpation of the adductor tendons or the insertion of the pubic bone or both; Groin pain during active adduction against resistance (squeeze test); Pain during adduction against resistance had to be less than six*, based on the visual analogue scale (VAS).
7. In addition, at least two of the following criteria had to be present: a clear history of groin pain and stiffness in the morning, cough induced or sneeze-induced groin pain, nocturnal groin pain or radiological evidence demonstrating osteitis pubis or pain at the symphysis pubis due to palpation.

Exclusion Criteria:

1. Receiving physical therapy or other conventional therapy in the past 6 months.
2. Absence in one of the pre- or post-test sessions.
3. Absence of more than two sessions in practice sessions.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-20 (Estimated); Primary Completion 2025-06-20 (Estimated); Study Completion 2025-11-20 (Estimated)

PRIMARY OUTCOMES:
EMG | From enrollment to the end of treatment at 12 weeks
  To record electromyographic activity of selected lumbo-pelvic muscles, the skin surface of the participants will be cleansed with alcohol pads and shaved to remove any hair in the designated area. Subsequently, to reduce skin electrical resistance, the skin will be lightly abraded with a soft sandpaper until its color visibly lightens. Surface electrodes, spaced 2 centimeters center-to-center along the muscle fibers, will then be affixed in the direction of the muscle fibers. The selected muscles for the lumbar region include the right rectus abdominis, internal oblique, and multifidus, while for the pelvic region, the iliocostalis lumborum and gluteus medius will be considered. Electrodes will be positioned according to SENIAM protocols for the respective muscles of interest. Proper electrode placement will be verified through manual assessment techniques, and electromyographic signals will be assessed and analyzed.
ESST | From enrollment to the end of treatment at 12 weeks
  The ESST was administered using a version standardized from previous literature. The units of measurement were changed from feet to meters, resulting in a slightly longer course of 4 m in length with four 1 m (3.28 ft) increments. The starting position was changed from the center cone to the far left cone in order to standardize the starting position, and each 1 m increment was marked with a strip of tape and a cone, which allowed for easier scoring of the test. The raters were positioned in front of and behind the participant. The participant began in a standing position behind the far left cone and was instructed not to cross his feet while sidestep ping. On the "go" command, the participant sidestepped to the right until his right foot had touched or crossed the outside cone or tape mark. The participant then side-stepped to the left until his left foot had touched or crossed the left outside cone or tape mark. The participant sidestepped back and forth to the outside cones as rapi
T-TEST | From enrollment to the end of treatment at 12 weeks
  The T-test was set up and administered using the protocol outlined by Semenick (1984). Upon the "Go" command, the sub- jects were instructed to sprint forward 9.10 m (10 yd), touch the cone with their right hand and without crossing their feet, side shuffle 4.55 m (5 yd) to the left, and touch the cone with their left hand. The subject then shuffles to the right 9.10 m (10 yd), touches the cone with their right hand, and returns to the center cone by side shuffling 4.55 m (5 yd). The subject then touches the center cone with their left hand and back pedals 9.10 m (10 yd) through the finish line, ensuring that balance is maintained. The intraclass reliability of the T-test was 0.98 across 3 trials in Pauole study (2000)(110) and 0.88 - 0.95 in Stewart study (2014)(111).
Y balance test | From enrollment to the end of treatment at 8 weeks
  YBT test performance was assessed with a Y Balance Test Kit. Before assessment, participants were acquainted with the Y-Balance Test (YBT) by practicing on their injured limb. The YBT was performed on a platform. Throughout the task, the standing leg remained on the platform, while the other leg executed error-free maximum reach in three directions: anterior, posteromedial, and posterolateral. Maximum distances in each direction, relative to the stance leg, were measured. During the test, participants kept their hands on their waists, and each direction was repeated three times with a 10-second rest between trials.
Groin Pain | From enrollment to the end of treatment at 12 weeks
  Pain was assessed and recorded based on the visual analogue scale (VAS) in the following two situations: (i) pain during the hip adduction against resistance (squeeze test) and (ii) pain during functional tests (the average earned from the two functional tests)(54).

IPD SHARING:
Plan to Share IPD: Yes
only IPD used in the results publication

REFERENCES:
- [Background] Yousefzadeh A, Shadmehr A, Olyaei GR, Naseri N, Khazaeipour Z. Effect of Holmich protocol exercise therapy on long-standing adductor-related groin pain in athletes: an objective evaluation. BMJ Open Sport Exerc Med. 2018 Jun 26;4(1):e000343. doi: 10.1136/bmjsem-2018-000343. eCollection 2018. PMID 30018787
- [Background] Tak I PhD, MScPT, Langhout R MMT PT, Bertrand B MScPT, Barendrecht M MPTS, Stubbe J PhD, Kerkhoffs G PhD, MD, Weir A PhD, MBBS. Manual therapy and early return to sport in football players with adductor-related groin pain: A prospective case series. Physiother Theory Pract. 2020 Sep;36(9):1009-1018. doi: 10.1080/09593985.2018.1531096. Epub 2018 Oct 11. PMID 30307775
- [Background] Jha S, Bajpai S, Mishra R. The Comparative Study between Active Physical Training versus Active Resistance Training in Groin Pain among Young Gymnasts. Central India Journal of Medical Research. 2023;2(01):8-12.
- [Background] Harris-Hayes M, Zorn P, Steger-May K, Buss J, Burgess MM, DeMargel RD, et al. Comparison of Joint Mobilization and Movement Pattern Training for Hip-related Groin Pain: Ancillary Analysis to Assess 12 Month Outcomes of a Pilot Randomized Clinical Trial. JOSPT Open. 2024;2(1):1-26.
- [Background] Delahunt E, Thorborg K, Khan KM, Robinson P, Holmich P, Weir A. Minimum reporting standards for clinical research on groin pain in athletes. Br J Sports Med. 2015 Jun;49(12):775-81. doi: 10.1136/bjsports-2015-094839. PMID 26031644
- [Background] Verrall GM, Slavotinek JP, Fon GT, Barnes PG. Outcome of conservative management of athletic chronic groin injury diagnosed as pubic bone stress injury. Am J Sports Med. 2007 Mar;35(3):467-74. doi: 10.1177/0363546506295180. Epub 2007 Jan 31. PMID 17267768
- [Background] Zeppieri G, Smith MS, Roach RP. Nonsurgical Management of Adductor-related groin pain with Ultrasound-Guided Platelet-Rich Plasma Injection and Physical Therapy in a Competitive Soccer Player: A Case Report. Int J Sports Phys Ther. 2024 Jul 1;19(7):898-909. doi: 10.26603/001c.120209. eCollection 2024. PMID 38966832
- [Background] Holmich P, Uhrskou P, Ulnits L, Kanstrup IL, Nielsen MB, Bjerg AM, Krogsgaard K. Effectiveness of active physical training as treatment for long-standing adductor-related groin pain in athletes: randomised trial. Lancet. 1999 Feb 6;353(9151):439-43. doi: 10.1016/S0140-6736(98)03340-6. PMID 9989713
- [Background] Holmich P. Long-standing groin pain in sportspeople falls into three primary patterns, a "clinical entity" approach: a prospective study of 207 patients. Br J Sports Med. 2007 Apr;41(4):247-52; discussion 252. doi: 10.1136/bjsm.2006.033373. Epub 2007 Jan 29. PMID 17261557